CLINICAL TRIAL: NCT05822024
Title: Promoting Pupils' Physical Literacy
Acronym: 3PL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Clinical Research and Prevention (Network)
Collaborators: University of Copenhagen (Other); TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Peter Bentsen, Center Director and Affiliated Professor, Center for Clinical Research and Prevention
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TRYG153181
Record Dates: First submitted 2023-04-03; First posted 2023-04-20 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Literacy
Keywords: Physical literacy; Physical education; School children; School based intervention; Education; Health promotion; Prevention
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Two schools (grade 4-5) will be randomly assigned to recieve the 3PL intervention in their physical education classes during one school year.
  Interventions: Behavioral: Promoting Pupils' Physical Literacy Intervention
- Control group (No Intervention): Two schools (grade 4-5) will be randomly assigned to the control group and will continue their normal physical education classes.

INTERVENTIONS:
Behavioral: Promoting Pupils' Physical Literacy Intervention — The physical literacy intervention 3PL is based on activities, games, and modifications of the physical education classes to target and enhance pupils' physical literacy.
  Other Names: 3PL
  Arms: Intervention group

SUMMARY:
This pilot study aims to test the feasibility and acceptability of a previously developed and tested physical literacy (PL) intervention. A promising and internationally tested intervention, the Youth Physical Activity Towards Health (Y PATH), is based on the theory of PL and has proven to be effectful on children's PA levels and motor skills The Promoting Pupils' Physical Literacy (3 PL) project aims to test the feasibility and acceptability of the previously developed and tested Y-PATH intervention in a Danish context among a pupils (9 11 years of age). The hypothesis is that a revised 3 PL intervention protocol, aiming to increase pupils' PL, is ready for effectiveness testing by the end of this project.

DETAILED DESCRIPTION:
This pilot study aims to test the feasibility and acceptability of a previously developed and tested physical literacy (PL) intervention. Regular participation in physical activity (PA) through life can improve health and reduce the risk of developing several chronic diseases like diabetes, cancer, and cardiovascular disease. However, a considerable number of Danish children and adolescents do not meet national PA recommendations. Over the last few years, the construct of PL has gained popularity around the world and has become recognized as a proximal measure for lifelong engagement in PA. PL is a multidisciplinary and comprehensive concept describing an individual's prerequisites to participate in and adhere to physical activities throughout the life course PL includes the elements motivation, confidence, motor skills, physical capacity, knowledge and understanding. In Denmark, development towards theoretically driven and evidence-based PL interventions that aim to increase children's PL have not yet begun. A promising and internationally tested intervention, the Youth Physical Activity Towards Health (Y-PATH), is based on the theory of PL and has proven to be effectful on children's PA levels and motor skills. The Promoting Pupils' Physical Literacy (3 PL) project aims to test the feasibility and acceptability of the previously developed and tested Y-PATH intervention in a Danish context among pupils (9-11 years of age). The hypothesis is that a revised 3 PL intervention protocol, aiming to increase pupils' PL, is ready for effectiveness testing by the end of this project.

Four schools will be recruited and randomly assigned to intervention or control condition. The primary outcomes include the feasibility and acceptability of the 3 PL intervention and will be in concordance with guidance proposed by the Medical Research Council and The Common Guidelines for Education Research and Development. Feasibility of the practicality and recruitment process will be assessed within a document log administered by the project group. The acceptability including demand and experiences, and the intervention implementation degree (secondary outcome) will be evaluated by short bimonthly questionnaires to teachers and interviews with pupils, teachers, parents, and school managers. Preliminary effectiveness (secondary outcome) will be tested by comparing changes in pupils' PL assessed with the Danish Assessment of Physical Literacy (DAPL) tool.

First and foremost, the testing of feasibility and acceptability of a previously developed international intervention will provide a revised 3 PL intervention, a Template for Intervention Description and Replication TIDieR checklist and a protocol, which will provide a solid empirical and theoretical foundation for a future upscaled effectiveness study. The development of a TIDieR checklist and a protocol provides international and national researchers the opportunity to use and compare effectiveness across countries and cultures.

ELIGIBILITY:
Inclusion Criteria:

School/class-level

* Non-special needs municipal school classes
* Classes that are not in other school development or research projects which would most likely influence and bias the results

Pupil-level

* Pupils with parents/guardians who have provided written informed consent, allowing their child to participate
* Pupils who have provide an oral assessment

Exclusion Criteria:

* Pupils who do not live up to the inclusion criteria

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 336 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Acceptance rate | 6 months
  Percentage of invited schools participating.
Success of intervention implementation in PE lessons | 11 months
  Three observations during physical education lessons (PE) that assess the acceptability of the intervention. Also, PE teachers will receive a weekly questionnaire to assess whether they have used the intervention materials in their PE lessons.
Success of intervention implementation in school systems | 11 months
  Qualitative interviews with school managers and teachers will be undertaken to detect perceived positive or negative effects on organization and how the intervention fits within the school culture.
Success of intervention implementation for pupils | 11 months
  Qualitative interviews with pupils will be undertaken to understand their experiences of the PE lessons.

SECONDARY OUTCOMES:
Physical literacy (preliminary effectiveness) | 11 months
  This study will assess PL among the pupils before and after the intervention period using the Danish Assessment of Physical Literacy (DAPL) that has been developed and validated in the DAPL project supported by TrygFonden #125640.
Daily physical activity (preliminary effectiveness) | 11 months
  Physical Activity will be measured with Axivity® AX3 accelerometers worn for 7 consecutive days. Axivity tracks physical activity in activity counts.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bentsen, PhD, Principal Investigator — Center for Clinical Research and Prevention; Peter Elsborg, PhD, Study Director — Center for Clinical Research and Prevention; Mads Bølling, PhD, Study Director — Center for Clinical Research and Prevention; Thea Toft Amholt, PhD, Study Director — Center for Clinical Research and Prevention; Glen Nielsen, PhD, Study Director — University of Copenhagen; Paulina Melby, PhD, Study Director — University of Copenhagen; Mette Kurtzhals, Cand.scient, Study Director — University of Southern Denmark
Locations (3):
- Denmark (3):
  - Center for Clinical Research and Prevension, Frederiksberg and Bispebjerg Hospital, Copenhagen, Frederiksberg
  - University of Copenhagen, Copenhagen, Nørrebro
  - University of Southern Denmark, Odense, Odense M

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Adaptation Protocol — https://osf.io/wd5ur/